CLINICAL TRIAL: NCT04548726
Title: Hemodynamic Matched Comparison of the Balloon-Expandable Transcatheter Heart Valves Myval and Sapien-3 for the Treatment of Aortic Stenosis
Acronym: MATCH-BALL
Status: Completed | Type: Observational
Sponsor: Ignacio J. Amat Santos (Other)
Responsible Party: Sponsor-Investigator, Ignacio J. Amat Santos, Coordinator of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Organization: Hospital Clínico Universitario de Valladolid (Other)
Other Study IDs: MATCH-BALL
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Regurgitation
Keywords: TAVI; TAVR; Balloon-Expandable transcatheter heart valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sapien 3: Patients with aortic stenosis treated with Sapien 3 (Edwards Lifesciences, Irvine, CA, USA) TAVI
  Interventions: Device: Sapien 3 Transcather Aortic Valve Implant
- Myval: Patients with aortic stenosis treated with Myval (Meril Life Sciences Pvt. Ltd., India) TAVI
  Interventions: Device: Myval Transcather Aortic Valve Implant

INTERVENTIONS:
Device: Sapien 3 Transcather Aortic Valve Implant — Implant of a Ballon Expandable Aortic Valve Sapien 3 (Edwards Lifesciences, Irvine, CA, USA) prosthesis via a transcatheter procedure.
  Groups: Sapien 3
Device: Myval Transcather Aortic Valve Implant — Implant of a Ballon Expandable Aortic Valve Myval (Meril Life Sciences Pvt. Ltd., India) prosthesis via a transcatheter procedure.
  Groups: Myval

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is recommended for patients with severe aortic stenosis (AS) at high to intermediate surgical risk. Despite similar mortality rates compared to surgical aortic valve replacement (SAVR) in this setting, the rate para-valvular leak (PVL) remains higher and has been associated to higher mortality even at mild degree. This is one of the major concerns to extend TAVI to low surgical risk, although the favorable results from PARTNER 3.

The presence of moderate to severe PVL after TAVI is associated to a 2- and 3- fold increase in the mortality rate at 30-day and 1-year follow-up, respectively (24-29).

Prosthesis-patient mismatch (PPM) adversely affects functional improvement and exercise tolerance, left ventricular (LV) mass regression, and late structural valve deterioration. Many studies have previously investigated PPM after surgical AVR suggesting the presence of this problem in more than 40% of the surgically treated patients. This rate was significantly lower with the balloon-expandable Sapien (Edwards Lifesciences, Irvine, California), with PPM that varied from 8% to 18%, but in both cases (patients harboring TAVI and those with SAVR) the mortality rate was higher in the presence of PPM.

Under the hypothesis that there are differences in terms of transvalvular gradients and residual para-valvular leak amongst different balloon-expandable TAVI devices available in the market, the aim of the MATCH-BALL study is to compare the hemodynamic performance of two balloon-expandable TAVI devices, Sapien 3 (Edwards Lifesciences, Irvine, CA, USA) and Myval (Meril Life Sciences Pvt. Ltd., India).

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with aortic stenosis (effective aortic<1.0 cm2) accepted for a TAVI procedure by the Heart Team.
* Implantation of Sapien-3 transfemoral valve or Myval transfemoral prosthesis.
* Availability of the variables selected for the matching process: Left ventricular ejection fraction, aortic annulus diameter and area, eccentricity index, and calcium score (all measured using computed tomography), body surface area, and body mass index.
* Availability of imaging studies at baseline and at discharge or 30-day follow up.

Exclusion Criteria:

* Failure to comply with matching criteria.
* Failure to properly analyse images in the echo core-lab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent TAVI with any of the previously explained self-expandable devices in the participating institutions and have at least one transthoracic echocardiography after TAVI procedure will be included. Main baseline and procedural characteristics as well as in-hospital outcomes will be drawn from the prospective database available at each institution.
  Echocardiographic exams will be centrally analysed by two independent operators blinded to the TAVI device and the clinical outcomes as well as to any clinical information of the patients.
  Subjects treated with each device will be matched with patients who had undergone transcatheter aortic valve implantation with the alternative devices and clinical and echocardiographic variables will be compared. The final matching will be performed by random sampling without replacement.
Sampling Method: Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Mean transvalvular gradients | 30 days
  Mean Gradients measured in doppler echography are calculated based on the mean velocity of the tracing. The velocities are converted to pressure gradients using the Bernoulli equation.
Aortic valve area | 30 days
  Echography measured Aortic valve area
Aortic valve perivalvular leak | 30 days
  Echography measured perivalvular leak
Aortic valve central leak | 30 days
  Echography measured central leak
Aortic valve global leak | 30 days
  Echography measured global leak

SECONDARY OUTCOMES:
Cardiovascular mortality rate | 30 days
All-cause mortality rate | 30 days
Myocardial infarction rate | 30 days
Bleeding complications rate | 30 days
Acute kidney injury rate | 30 days
Vascular complications rate | 30 days
Conduction disorder rate | 30 days
Re-hospitalization rate | 30 days
Need for permanent pacemaker rate | 30 days
New York Heart Association (NYHA) functional class | 30 days

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (4):
  - Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Policlinico San Donato, San Donato Milanese
  - Ospedale San Raffaele, Segrate
- Spain (2):
  - Hospital Universitario de Gran Canaria Dr Negrin, Las Palmas de Gran Canaria
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No